CLINICAL TRIAL: NCT06636461
Title: Assessment of Dimensional Changes Following Grafting With Microfragmented Adipose Tissue Loaded on Allograft on Ridge Preservation Versus Allograft Only for Subsequent Implant Placement in the Maxillary Posterior Region, a Randomized Clinical Trial
Brief Title: Assessment of Dimensional Changes Following Grafting With Microfragmented Adipose Tissue Loaded on Allograft on Ridge Preservation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Omar Salem Alnahdi, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Assessment of dimensional chan
Record Dates: First submitted 2024-09-02; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hopeless Tooth
Keywords: hopeless tooth lesion or affected periodontium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microfragmented adipose tissue (Experimental): microfragmented adipose tissue loaded on allograft on ridge preservation
  Interventions: Procedure: microfragmented adipose tissue loaded on allograft
- allograft (Active Comparator): allograft only on ridge preservation
  Interventions: Procedure: microfragmented adipose tissue loaded on allograft

INTERVENTIONS:
Procedure: microfragmented adipose tissue loaded on allograft — microfragmented adipose tissue loaded on allograft on ridge preservation

SUMMARY:
Evaluation of maxillary alveolar ridge changes (bone quantity and quality as revealed by radiographic and Histomorphometry ) utilizing microfragmented adipose tissue loaded on allograft versus allograft only for maxillary posterior ridge preservation

DETAILED DESCRIPTION:
All patients involved in this study will be divided into two groups; each group will receive a different graft of bone augmentation: Adipose tissue loaded on allograft will be utilized for the study group and allograft only for the control group.

After 3-6 months, assessment of dimensional changes ( RG height & width) on CBCT is performed and Histomorphometry will be evaluated via core biopsy at the time of implant placement in both groups.

Radiographic assessment that will be achieved by CBCT scan will be used to calculate the changes of bone height and width from base line (1week) to 3-6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring implant treatment after tooth extraction due to either unrestorable caries lesions or affected periodontium.

Age group: above 18 years

• Remaining natural teeth have good periodontal tissue support and occlusion showed sufficient inter arch space for future prosthesis.

Exclusion Criteria:

* • General contraindications to implant surgery.

  * Subjected to irradiation in the head and neck area less than 1 year before implantation.
  * Poor oral hygiene and motivation.
  * Severe bruxism or clenching.
  * Systemic, immunologic or debilitating diseases that could affect normal bone healing & local pathosis.
  * Treated or under treatment of intravenous amino-bisphosphonates.
  * Active infection or severe inflammation in the area intended for implant placement.
  * Patients participating in other studies, if the present protocol could not be properly followed.
  * Heavy somkers

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge hight (bone quantity ) | Alveolar ridge hight (bone quantity ) by CBCT after 3-6 months
  By CBCT

SECONDARY OUTCOMES:
Alveolar ridge width. | Alveolar ridge width. by CBCT after 3-6 months
  By CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Universty, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All patients involved in this study will be divided into two groups; each group will receive a different graft of bone augmentation: Adipose tissue loaded on allograft will be utilized for the study group and allograft only for the control group.
  For both groups: All Patients of both groups will be evaluated radiographically immediately and after 3- 6 months post-operative by cone beam CT scan to record Alveolar ridge height and width.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After 6 months, patients will be evaluated histomorphometrically via core biopsy at the time of implant placement and radiographically via assessment of ridge height on CBCT.
  Radiographic assessment that will be achieved by CBCT scan will be used to calculate the changes of bone height and width from base line (1week) to 6 months postoperatively.